CLINICAL TRIAL: NCT06495060
Title: The Correlation Between Psychological Capital, Intention to Leave, Work Job and Environment Satisfaction, and Political Skills Among Different Generations Nurses
Status: Completed | Type: Observational
Sponsor: Mackay Memorial Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: 24MMHIS126e
Record Dates: First submitted 2024-06-30; First posted 2024-07-10 (Actual); Last update posted 2025-09-25 (Actual); Status verified 2024-07

CONDITIONS: Generation Gap
Keywords: Generation Nurses; Psychological Capital; Intention to leave

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (2):
- Clinical Nurse (Registered Nurse)
  Interventions: Other: No intervention (Only observation)
- Nursing Practitioners
  Interventions: Other: No intervention (Only observation)

INTERVENTIONS:
Other: No intervention (Only observation) — No intervention

SUMMARY:
Purpose

1. To understand the current status of demographic characteristics, inclination to resign, Psychological Capital, work environment and job satisfaction, and political skills among incumbent clinical nursing staff across different generations.
2. To understand the correlation and interaction between demographic characteristics, inclination to resign, Psychological Capital, work environment and job satisfaction, and political skills among incumbent clinical nursing staff across different generations.

Expected outcomes

1. This study will provide objective and empirical data on the psychological capital, turnover intention, work environment and satisfaction, and political skills of clinical nursing personnel from different generations. By examining demographic variables, further exploration of the correlations among different attributes such as units, age, and positions (e.g., clinical nurses, nursing supervisors, specialist nurses) can be conducted. Through the research findings, the current status and needs of clinical nursing can be understood.
2. The results of this study will enable clinical nursing units in the future to implement measures to improve the psychological capital and address turnover intentions of nursing personnel from different generations and positions. Based on this objective and concrete data, relevant courses or training programs can be developed to retain excellent clinical nursing personnel.

ELIGIBILITY:
Inclusion Criteria:

* Aged 20 years or older.
* Currently employed in a hospital and possessing a nursing license.
* Willing to participate in this study.
* Currently employed as full-time or part-time nursing staff at the hospital.

Exclusion Criteria:

* Nursing staff who do not possess a nursing license.
* Nursing staff who are unwilling to participate in the study.
* Nursing staff who have already completed the related research questionnaire in the pilot study.

Ages: 20 Years to 99 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Licensed nursing staff.
Sampling Method: Non-Probability Sample
Enrollment: 646 (Actual)
Dates: Start 2024-08-09 (Actual); Primary Completion 2025-04-03 (Actual); Study Completion 2025-05-08 (Actual)

PRIMARY OUTCOMES:
Psychological Capital | Baseline
  This study utilized the Psychological Capital Questionnaire (PCQ) developed by scholars Luthans. It is used to measure nurses' level of psychological capital. The PCQ consists of 24 items designed to assess the level of psychological capital among nursing staff. The subscales include:Self-Efficacy Scale, Hope Scale, Resilience Scale and Optimism Scale.
  The PCQ uses a 6-point Likert scale for scoring:
  1 = Strongly Disagree,2 = Disagree, 3 = Somewhat Disagree, 4 = Somewhat Agree, 5 = Agree, 6 = Strongly Agree.

SECONDARY OUTCOMES:
Intention to leave | Baseline
  The intention to leave scale was used to measure the frequency of nursing staff's thoughts about resigning. This single-item measure assessed oncology nurses' subjective perception of how often they had thoughts of quitting over the past week. The frequency was scored on a 1 to 5 scale:
  1 = Never, 2 = Rarely, 3 = Sometimes, 4 = Often, 5 = Always.
Political skill | Baseline
  The Political Skill Inventory (PSI) was used to measure the level of social skills among nursing staff. This scale includes four dimensions: Social Astuteness, Networking Ability, Interpersonal Influence, Apparent Sincerity
  The PSI uses a 5-point Likert scale for scoring:
  1 = Strongly Disagree, 2 = Mostly Disagree, 3 = Neutral, 4 = Mostly Agree, 5 = Strongly Agree.
self-actualization (Work Environment and Job Satisfaction Scale) | Baseline
  The Work Environment and Job Satisfaction Scale, developed by scholars Rossberg et al., was used to measure the sense of self-actualization among nursing staff. This scale consists of 10 items designed to evaluate nursing staff's perceptions of their work environment. The subscales include:Self-actualization, Workload, Conflict, Stress,
  The scale uses a 5-point Likert scale for scoring:
  1 = Not at all, 2 = Rarely, 3 = Sometimes, 4 = Often, 5 = Always

CONTACTS AND LOCATIONS:
Locations (1):
- Mackay Memorial Hospital, Taipei, Taiwan

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Aiken LH, Sloane DM. Nurses matter: more evidence. BMJ Qual Saf. 2020 Jan;29(1):1-3. doi: 10.1136/bmjqs-2019-009732. Epub 2019 Sep 9. No abstract available. PMID 31501231
- [Background] Al Maqbali M. Sleep disturbance among frontline nurses during the COVID-19 pandemic. Sleep Biol Rhythms. 2021;19(4):467-473. doi: 10.1007/s41105-021-00337-6. Epub 2021 Jul 1. PMID 34230810
- [Background] Rossberg JI, Eiring O, Friis S. Work environment and job satisfaction. A psychometric evaluation of the Working Environment Scale-10. Soc Psychiatry Psychiatr Epidemiol. 2004 Jul;39(7):576-80. doi: 10.1007/s00127-004-0791-z. PMID 15243696
- [Background] Luthans, F. (2002). The need for and meaning of positive organizational behavior. Journal of Organizational Behavior: The International Journal of Industrial, Occupational and Organizational Psychology and Behavior, 23(6), 695-706.
- [Background] Luthans, F., Avolio, B. J., Avey, J. B., & Norman, S. M. (2007). Positive psychological capital: Measurement and relationship with performance and satisfaction.
- [Background] Taggar, S., & Brown, T. C. (2001). Problem-solving team behaviors: Development and validation of BOS and a hierarchical factor structure. Small group research, 32(6), 698-726.
- [Background] Arslan, A., Ahokangas, P., Haapanen, L., Golgeci, I., Tarba, S. Y., & Bazel-Shoham, O. (2022). Generational differences in organizational leaders: an interpretive phenomenological analysis of work meaningfulness in the Nordic high-tech organizations. Technological Forecasting and Social Change, 180, 121717.
- [Background] Bae SH, Cho M, Kim O, Pang Y, Cha C, Jung H, Kim S, Jeong H. Predictors of actual turnover among nurses working in Korean hospitals: A nationwide longitudinal survey study. J Nurs Manag. 2021 Oct;29(7):2102-2114. doi: 10.1111/jonm.13347. Epub 2021 May 11. PMID 33894028
- [Background] Sinclair HA, Hamill C. Does vicarious traumatisation affect oncology nurses? A literature review. Eur J Oncol Nurs. 2007 Sep;11(4):348-56. doi: 10.1016/j.ejon.2007.02.007. Epub 2007 May 7. PMID 17482879
- [Background] Bautista JR, Lauria PAS, Contreras MCS, Maranion MMG, Villanueva HH, Sumaguingsing RC, Abeleda RD. Specific stressors relate to nurses' job satisfaction, perceived quality of care, and turnover intention. Int J Nurs Pract. 2020 Feb;26(1):e12774. doi: 10.1111/ijn.12774. Epub 2019 Aug 19. PMID 31423700
- [Background] Blanco-Donoso LM, Moreno-Jimenez J, Amutio A, Gallego-Alberto L, Moreno-Jimenez B, Garrosa E. Stressors, Job Resources, Fear of Contagion, and Secondary Traumatic Stress Among Nursing Home Workers in Face of the COVID-19: The Case of Spain. J Appl Gerontol. 2021 Mar;40(3):244-256. doi: 10.1177/0733464820964153. Epub 2020 Oct 7. PMID 33025850
- [Background] Boamah SA, Laschinger H. The influence of areas of worklife fit and work-life interference on burnout and turnover intentions among new graduate nurses. J Nurs Manag. 2016 Mar;24(2):E164-74. doi: 10.1111/jonm.12318. Epub 2015 Jun 30. PMID 26122304
- [Background] Burhanuddin, N. A. N., Ahmad, N. A., Said, R. R., & Asimiran, S. (2019). A systematic review of the psychological capital (PsyCap) research development: Implementation and gaps. International Journal of Academic Research in Progressive Education and Development, 8(3), 133-150.
- [Background] Chen H, Sun L, Du Z, Zhao L, Wang L. A cross-sectional study of mental health status and self-psychological adjustment in nurses who supported Wuhan for fighting against the COVID-19. J Clin Nurs. 2020 Nov;29(21-22):4161-4170. doi: 10.1111/jocn.15444. Epub 2020 Sep 1. PMID 32757428
- [Background] Christensen SS, Wilson BL, Edelman LS. Can I relate? A review and guide for nurse managers in leading generations. J Nurs Manag. 2018 Sep;26(6):689-695. doi: 10.1111/jonm.12601. Epub 2018 Jan 30. PMID 29380917
- [Background] Dewanto A, Wardhani V. Nurse turnover and perceived causes and consequences: a preliminary study at private hospitals in Indonesia. BMC Nurs. 2018 Dec 19;17(Suppl 2):52. doi: 10.1186/s12912-018-0317-8. eCollection 2018. PMID 30574016
- [Background] Dobnik M, Maletic M, Skela-Savic B. Work-Related Stress Factors in Nurses at Slovenian Hospitals - A Cross-sectional Study. Zdr Varst. 2018 Oct 1;57(4):192-200. doi: 10.2478/sjph-2018-0024. eCollection 2018 Dec. PMID 30294360
- [Background] Flinkman M, Salantera S. Early career experiences and perceptions - a qualitative exploration of the turnover of young registered nurses and intention to leave the nursing profession in Finland. J Nurs Manag. 2015 Nov;23(8):1050-7. doi: 10.1111/jonm.12251. Epub 2014 Sep 3. PMID 25186284
- [Background] Frey R, Robinson J, Wong C, Gott M. Burnout, compassion fatigue and psychological capital: Findings from a survey of nurses delivering palliative care. Appl Nurs Res. 2018 Oct;43:1-9. doi: 10.1016/j.apnr.2018.06.003. Epub 2018 Jun 18. PMID 30220354
- [Background] Hampton D, Welsh D. Work Values of Generation Z Nurses. J Nurs Adm. 2019 Oct;49(10):480-486. doi: 10.1097/NNA.0000000000000791. PMID 31517755
- [Background] Holtzhausen, J. D. V., Coetzee, S. K., & Ellis, S. M. (2020). Influence of the practice environment on community service nurses' subjective well-being, compassion practice and psychological capital. International Journal of Africa Nursing Sciences, 13, 100243.
- [Background] Joo, B.-K., Lim, D. H., & Kim, S. (2016). Enhancing work engagement: The roles of psychological capital, authentic leadership, and work empowerment. Leadership & Organization Development Journal, 37(8), 1117-1134.
- [Background] Karatepe, O. M., & Karadas, G. (2015). Do psychological capital and work engagement foster frontline employees' satisfaction? A study in the hotel industry. International Journal of Contemporary Hospitality Management, 27(6), 1254-1278.
- [Background] Koppel J, Deline M, Virkstis K. The Case for Focusing on Millennial Retention. J Nurs Adm. 2017 Jul/Aug;47(7-8):361-363. doi: 10.1097/NNA.0000000000000495. PMID 28727620
- [Background] Laschinger, H. K. S., & Fida, R. (2014). New nurses burnout and workplace wellbeing: The influence of authentic leadership and psychological capital. Burnout research, 1(1), 19-28.
- [Background] Luthans, F., Avolio, B. J., Avey, J. B., & Norman, S. M. (2007). Positive psychological capital: Measurement and relationship with performance and satisfaction. Personnel psychology, 60(3), 541-572.
- [Background] Rudolph CW, Rauvola RS, Costanza DP, Zacher H. Generations and Generational Differences: Debunking Myths in Organizational Science and Practice and Paving New Paths Forward. J Bus Psychol. 2021;36(6):945-967. doi: 10.1007/s10869-020-09715-2. Epub 2020 Sep 4. PMID 32901173
- [Background] Shapiro D, Duquette CE, Zangerle C, Pearl A, Campbell T. The Seniority Swoop: Young Nurse Burnout, Violence, and Turnover Intention in an 11-Hospital Sample. Nurs Adm Q. 2022 Jan-Mar 01;46(1):60-71. doi: 10.1097/NAQ.0000000000000502. PMID 34860802
- [Background] Spreitzer, G. M. (1995). Psychological empowerment in the workplace: Dimensions, measurement, and validation. Academy of management Journal, 38(5), 1442- 1465.
- [Background] Sweet, J., & Swayze, S. (2017). The multi-generational nursing workforce: Analysis of psychological capital by generation and shift. Journal of Organizational Psychology, 17(4).
- [Background] Tan SHE, Chin GF. Generational effect on nurses' work values, engagement, and satisfaction in an acute hospital. BMC Nurs. 2023 Mar 30;22(1):88. doi: 10.1186/s12912-023-01256-2. PMID 36997911
- [Background] Ting, H., Lim, T.-Y., de Run, E. C., Koh, H., & Sahdan, M. (2018). Are we baby boomers, gen X and gen Y? A qualitative inquiry into generation cohorts in Malaysia. Kasetsart Journal of Social Sciences, 39(1), 109-115.
- [Background] Viseu, J., de Jesus, S. N., Rus, C., & Canavarro, J. M. (2016). Teacher motivation, work satisfaction, and positive psychological capital: A literature review. Electronic Journal of Research in Education Psychology, 14(39), 439-461.
- [Background] Waltz LA, Munoz L, Weber Johnson H, Rodriguez T. Exploring job satisfaction and workplace engagement in millennial nurses. J Nurs Manag. 2020 Apr;28(3):673-681. doi: 10.1111/jonm.12981. Epub 2020 Apr 6. PMID 32068932
- [Background] Wang X, Liu L, Zou F, Hao J, Wu H. Associations of Occupational Stressors, Perceived Organizational Support, and Psychological Capital with Work Engagement among Chinese Female Nurses. Biomed Res Int. 2017;2017:5284628. doi: 10.1155/2017/5284628. Epub 2017 Jan 12. PMID 28168198
- [Background] Wang Y, Chang Y, Fu J, Wang L. Work-family conflict and burnout among Chinese female nurses: the mediating effect of psychological capital. BMC Public Health. 2012 Oct 29;12:915. doi: 10.1186/1471-2458-12-915. PMID 23107113
- [Background] Yan D, Wen F, Li X, Zhang Y. The relationship between psychological capital and innovation behaviour in Chinese nurses. J Nurs Manag. 2020 Apr;28(3):471-479. doi: 10.1111/jonm.12926. Epub 2020 Apr 20. PMID 31811781
- [Background] Zamanzadeh V, Valizadeh L, Khajehgoodari M, Bagheriyeh F. Nurses' experiences during the COVID-19 pandemic in Iran: a qualitative study. BMC Nurs. 2021 Oct 14;20:198. doi: 10.1186/s12912-021-00722-z. eCollection 2021. PMID 34649547